CLINICAL TRIAL: NCT02803203
Title: A Phase 1/2 Study of Combination Osimertinib and Bevacizumab as Treatment for Patients With EGFR-mutant Lung Cancers
Brief Title: Osimertinib and Bevacizumab as Treatment for EGFR-mutant Lung Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-033
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-03

CONDITIONS: Non-small Cell Lung Cancer; EGFR-mutant Lung Cancers
Keywords: Osimertinib; bevacizumab; metastatic; 16-033
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — osimertinib; Bevacizumab

ARMS (1):
- osimertinib and bevacizumab (Experimental): Phase 1:
  3+3 dose escalation design 2 dose levels Dose level -1: Osimertinib 40mg daily Maximum accrual = 12 Bevacizumab 15mg/kg q3 weeks Dose level 1: Osimertinib 80mg daily Bevacizumab 15mg/kg q3 Weeks
  Phase 2:
  Use MTD determined during phase 1
  Interventions: Drug: osimertinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: osimertinib
  Other Names: AZD9291
Drug: Bevacizumab

SUMMARY:
The purpose of this study is to test the safety of combining the drugs osimertinib and bevacizumab at different dose levels. The investigators want to find out what effects, good and/or bad, taking osimertinib and bevacizumab has on the patient and lung cancer. This study will try to find the best dose of osimertinib and bevacizumab given together that does not cause significant side effects. Once the investigators determine that combining osimertinib and bevacizumab is safe, they want to see if the combination is effective in treating lung cancers with the EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Advanced biopsy-proven metastatic non-small cell lung cancer
* Somatic activating mutation in EGFR
* No prior treatment with an EGFR TKI
* No prior treatment with a VEGF inhibitor
* Measurable (RECIST 1.1) indicator lesion not previously irradiated
* Karnofsky performance status (KPS) ≥ 70%
* Age >18 years old
* Adequate organ function

  * AST, ALT ≤ 3 x ULN
  * Total bilirubin ≤ 1.5x ULN
  * Creatinine ≤ 1.5x ULN OR calculated creatinine clearance > 60ml/min
  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
  * Hemoglobin≥8.0 g/dL
  * Platelets ≥100,000/mm3

Exclusion Criteria:

* Any contra-indications to bevacizumab which include but are not limited to recent

  1. Any previous venous thromboembolism > NCI CTCAE Grade 3
  2. Severe uncontrolled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥ 100mmHg)
  3. Cardiovascular disease including stroke of myocardial infarction <6 months prior to study enrollment, New York Heart Association Grade 2 or greater congestive heart failure, serious cardiac arrythmia uncontrolled by medication
  4. Hemorrhagic brain metastases. Asymptomatic (not requiring escalating doses of steroids) brain metastases are acceptable.
  5. History of severe proteinuria (urine dipstick ≥ 2+ or 24 hr urine > 2gm/24hr)
  6. Prior history of hypertensive crisis or hypertensive encephalopathy
  7. History of a central nervous system disease (e.g. seizures) unrelated to cancer unless adequately treated with standard medical therapy
  8. Significant vascular disease (e.g. aortic aneurysm requiring surgical repair)≥ 6 months prior to study enrollment
  9. History of hemoptysis (≥1/2 teaspoon of bright red blood per episode) within the last 3 months
  10. Evidence of a bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
  11. Current or recent (within 10 days of study drug start) use of aspirin (>325mg daily), clopidogrel (>75mg daily).
  12. Recent initiation of full dose oral or parental anticoagulants that have not been in place for at least 2 weeks.
  13. Tumor invading or abutting major blood vessels
  14. Tumor histology classified by squamous cell histology.
  15. Any history of abdominal fistula or GI perforation within 6 months of study enrollment
* Pregnant or lactating women
* Any type of systemic anticancer therapy (chemotherapy or experimental drugs) within 2 weeks of starting treatment on protocol
* Any radiotherapy within 1 week of starting treatment on protocol
* Any major surgery within 4 weeks of starting treatment on protocol
* Any evidence of clinically significant interstitial lung disease
* Known hypersensitivity to any component of bevacizumab and osimertinib

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Yu HA, Schoenfeld AJ, Makhnin A, Kim R, Rizvi H, Tsui D, Falcon C, Houck-Loomis B, Meng F, Yang JL, Tobi Y, Heller G, Ahn L, Hayes SA, Young RJ, Arcila ME, Berger M, Chaft JE, Ladanyi M, Riely GJ, Kris MG. Effect of Osimertinib and Bevacizumab on Progression-Free Survival for Patients With Metastatic EGFR-Mutant Lung Cancers: A Phase 1/2 Single-Group Open-Label Trial. JAMA Oncol. 2020 Jul 1;6(7):1048-1054. doi: 10.1001/jamaoncol.2020.1260. PMID 32463456
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Osimertinib and Bevacizumab: Phases 1+2: Osimertinib + Bevacizumab 80 mg Osimertinib PO QD and 15 mg/kg Bevacizumab IV Q3W
  This section accurately reflects the flow of participants as all participants were enrolled into the same dosing cohort. This protocol utilized a dose de-escalation model where the initial dose was continued for Phase 2.
Period: Overall Study
Arm/Group | Osimertinib and Bevacizumab
Started | 49
Completed | 0
Not Completed | 49
Not completed — Adverse Event | 4
Not completed — Death | 4
Not completed — Progressive disease | 29
Not completed — Withdrawal by Subject | 8
Not completed — Complete resection of target disease | 2
Not completed — Switched to commercial Osi | 1
Not completed — Participant moved away | 1

BASELINE CHARACTERISTICS:
Arm/Group | Osimertinib and Bevacizumab
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Osimertinib Maximum Tolerated Dose (MTD) (Phase I)
Description: The MTD (maximum tolerated dose)/recommended phase 2 dose will be the highest dose level at which <1 DLT is detected in the first cycle for 6 treated patients. If only 3 patients are treated at a dose level being considered for the MTD, an additional 3 patients will be enrolled.
Time Frame: 1 year
Measure: Number; unit: mg
Groups:
- Osimertinib and Bevacizumab: Phase 1 participants
Arm/Group | Osimertinib and Bevacizumab
Number analyzed (Participants) | 6
mg | 80

2. Primary Outcome: Bevacizumab Maximum Tolerated Dose (MTD) (Phase I)
Description: as for outcome 1
Time Frame: 1 year
Measure: Number; unit: mg/kg
Arm/Group | Osimertinib and Bevacizumab
Number analyzed (Participants) | 6
mg/kg | 15

3. Primary Outcome: Progression-free Survival (Phase II)
Description: Tumor response will be assessed using RECIST 1.1. A CT chest/abdomen/pelvis will be performed to demonstrate all known areas of measurable disease. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib and Bevacizumab
Number analyzed (Participants) | 49
Participants
  Confirmed Partial Response/PR | 34
  Unconfirmed Partial Response/PR | 5
  Stable Disease/SD | 9
  Not Evaluable/NE | 1

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Osimertinib and Bevacizumab: Phases 1+2: Osimertinib + Bevacizumab 80 mg Osimertinib PO QD and 15 mg/kg Bevacizumab IV Q3W
  This section accurately reflects the flow of participants as all participants were enrolled into the same dosing cohort.
Arm/Group | Osimertinib and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 37/49
Serious Adverse Events (participants affected / at risk) | 26/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib and Bevacizumab (N=49)
Sinus tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Cholangitis (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Fever (General disorders) | 4
Non-cardiac chest pain (General disorders) | 3
Sudden death NOS (General disorders) | 1
Infections and infestations - Other, specify: Thyroid Gland (Infections and infestations) | 1
Lung infection (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 3
Confusion (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Dizziness (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Vascular disorders - Other (Vascular disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib and Bevacizumab (N=49)
Alanine aminotransferase increased (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3
CPK increased (Investigations) | 19
Diarrhea (Gastrointestinal disorders) | 49
Dizziness (Nervous system disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 23
Dysgeusia (Nervous system disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Edema limbs (General disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19
Fatigue (General disorders) | 40
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gen disorders & admin site conditions Other (General disorders) | 22
Headache (Nervous system disorders) | 5
Hematuria (Renal and urinary disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 12
Hypertension (Vascular disorders) | 49
Hyponatremia (Metabolism and nutrition disorders) | 3
Lymphocyte count decreased (Investigations) | 49
Mucositis oral (Gastrointestinal disorders) | 40
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Myositis (Musculoskeletal and connective tissue disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
Nausea (Gastrointestinal disorders) | 27
Neutrophil count decreased (Investigations) | 8
Paresthesia (Nervous system disorders) | 3
Paronychia (Infections and infestations) | 16
Platelet count decreased (Investigations) | 49
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Proteinuria (Renal and urinary disorders) | 49
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 33
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 26
Skin & subcutaneous tissue disorders Other (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 4
Vomiting (Gastrointestinal disorders) | 8
Weight loss (Investigations) | 12
White blood cell decreased (Investigations) | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT02803203/Prot_SAP_000.pdf